CLINICAL TRIAL: NCT01501864
Title: School Support as Structural HIV Prevention for Adolescent Orphans in Kenya
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Moi University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIRE-0580; R01MH092215 (NIH)
Record Dates: First submitted 2011-11-03; First posted 2011-12-30 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: HIV
Keywords: HIV prevention; HSV-2; Schooling; Kenya; Orphans; School support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- School Support Group (Experimental): School Support Intervention
  Interventions: Behavioral: School Support Intervention
- Control (No Intervention): No school support

INTERVENTIONS:
Behavioral: School Support Intervention — Comprehensive school support is provided that includes payment of school fees, school uniform, and a nurse researcher who monitors attendance and addresses problems that may lead to school absence and dropout.
  Arms: School Support Group

SUMMARY:
The purpose of this study is to test whether school support can keep adolescent Kenyan orphans in school, reduce sexual risk behaviors, and prevent HIV /HSV-2 infection.

DETAILED DESCRIPTION:
This study examines the impact of school support as a structural intervention, tested among adolescent orphans in Siaya District, Nyanza Province, Kenya.

Aims for the proposed study are: 1) To experimentally test whether providing comprehensive school support to Kenyan orphaned boys and girls will reduce school dropout, reduce sexual risk behaviors, and prevent HIV/HSV-2 infection; 2) To conduct a process evaluation of the implementation of the program; and 3) To conduct comparative cost effectiveness analyses, specifying the intervention's cost and return on investment as evidenced by cost per unit improvement in the primary outcomes of school enrollment, delay of sexual debut and prevention of risk behaviors and HIV/HSV-2 infection, as well as by gains in health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Orphan (one or both parents deceased)
* In Grade 7 or 8 in a primary school participating in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Dropped out of school | From date of randomization until drop out from school, up to 3 years
Change from baseline in ever had sexual intercourse at 1 year | Baseline and 1 year
Change from baseline in ever had sexual intercourse at 2 years | Baseline and 2 years
Change from baseline in ever had sexual intercourse at 3 years | Baseline and 3 years
HIV Incidence | 3 years
HSV-2 Incidence | 3 years

SECONDARY OUTCOMES:
Ever married or ever pregnant | From date of randomization until marriage or preganancy, up to 3 years
Health-related quality of life | Baseline and 1 year
Health-related quality of life | Baseline and 2 years
Health-related quality of life | Baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyunsan Cho, Ph.D., Principal Investigator — Pacific Institute for Research and Evaluation
Locations (2):
- Pacific Institute for Research and Evaluation, Chapel Hill, North Carolina, United States
- Moi University, Department of Nursing Sciences, Eldoret, Kenya

REFERENCES:
- [Derived] Cho H, Mbai I, Luseno WK, Hobbs M, Halpern C, Hallfors DD. School Support as Structural HIV Prevention for Adolescent Orphans in Western Kenya. J Adolesc Health. 2018 Jan;62(1):44-51. doi: 10.1016/j.jadohealth.2017.07.015. Epub 2017 Nov 6. PMID 29107569
- [Derived] Hallfors DD, Cho H, Mbai II, Millimo BW, Atieno C, Okumu D, Luseno WK, Hartman S, Halpern CT, Hobbs MM. Disclosure of HSV-2 serological test results in the context of an adolescent HIV prevention trial in Kenya. Sex Transm Infect. 2015 Sep;91(6):395-400. doi: 10.1136/sextrans-2015-052025. Epub 2015 Jul 2. PMID 26139208
- [Derived] Cho H, Luseno W, Halpern C, Zhang L, Mbai I, Milimo B, Hallfors DD. Discordance of HIV and HSV-2 biomarkers and self-reported sexual behaviour among orphan adolescents in Western Kenya. Sex Transm Infect. 2015 Jun;91(4):260-5. doi: 10.1136/sextrans-2014-051720. Epub 2014 Nov 6. PMID 25378660